CLINICAL TRIAL: NCT02117804
Title: Validating Discharge Planning Decision Support in a Regional Community Hospital
Brief Title: Early Screen for Discharge Planning in Community Hospitals
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Diane Holland, Clinical Nurse Researcher, Mayo Clinic
Other Study IDs: 14-002495
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Hospitalization
Keywords: Discharge Planning; Decision Support
MeSH Terms: interventions — Patient Discharge

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High ESDP Score: Patients with 10 or greater score on the Early Screen for Discharge Planning at the time of admission.
  Interventions: Other: Early Screen for Discharge Planning
- Low ESDP Score: Patients with 9 or lower score on the Early Screen for Discharge Planning at the time of admission.
  Interventions: Other: Early Screen for Discharge Planning

INTERVENTIONS:
Other: Early Screen for Discharge Planning — This screen is completed by a study coordinator within 24 hours of patient admission to the hospital. The screen measures four variables available from routine hospital admission clinical data (walking limitation, age, living alone prior to admission, and level of disability) that exhibit high sensitivity and specificity (AUC's were .82 and.84) in identifying patients who should receive targeted attention from a DP expert.

SUMMARY:
The purpose of this study is to determine the predictive performance of the Early Screen for Discharge Planning (ESDP) tool in a regional community hospital. The central hypothesis is that the ESDP differentiates between patients in a regional community hospital who would benefit from those who would not benefit from early discharge-planning intervention as measured by problems and unmet continuing care needs, quality of life, length of stay, and referrals to post-acute services.

DETAILED DESCRIPTION:
Patients who are hospitalized for medical or surgical reasons who consent to the study will be screened within 24 hours of hospital admission using the Early Screen for Discharge Planning (ESDP). The ESDP is a four-item screening tool used to determine on admission which patients are likely to have complex discharge plans and could benefit from early engagement of discharge planning personnel. The ESDP yields a total score, and those with a score of 10 or greater are considered to have a "high score" and likely to have a complex discharge plan. Those with a score of 9 or below have a "low score". The ESDP screen has been proven to be valid in large academic medical centers. This study will determine if the screen performs with the same validity in a small community hospital.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Able to read and speak English
* Returning home in the community after discharge

Exclusion Criteria:

* Discharged to facility care
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study targets adults hospitalized for a variety of medical and surgical conditions in a rural regional community hospital that is part of a large health system in the Midwest. The sample will be limited to adults who are returning home in the community, because the investigators are primarily interested in the problems and unmet needs encountered after discharge during the recovery period at home. To enhance the generalizability of the results, the sample will be stratified based on 2010 national estimates of age categories for hospitalized adults.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of problems reported after discharge, measured by the Problems After Discharge Questionnaire - English Version (PADQ-E) | 1 week after hospital discharge
  A problem is defined as any worry, limitation, concern, or difficulty reported by the patient. The Problems After Discharge Questionnaire - English Version measures important patient factors often overlooked that contribute to poor post-acute recovery experience which are recognized as important factors likely to impact readmission.

SECONDARY OUTCOMES:
Number of unmet needs reported after discharge, measured by the Problems After Discharge Questionnaire - English Version (PADQ-E) | 1 week after hospital discharge
  An unmet need is a need for help identified by the patient that is reported to be inadequately met. The Problems After Discharge Questionnaire - English Version measures important patient factors often overlooked that contribute to poor post-acute recovery experience which are recognized as important factors likely to impact readmission.
Quality of life, measured by the EuroQoL-5D | 1 week after hospital discharge
  The EuroQoL-5D (EQ-5D) is a standardized instrument for use as a measure of health out-come. Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status that can be used in the clinical and economic evaluation of health care.

CONTACTS AND LOCATIONS:
Overall Officials: Diane E. Holland, PhD, RN, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Health System - Eau Claire, Eau Claire, Wisconsin, United States